CLINICAL TRIAL: NCT05245942
Title: Monitoring of the Safety and the Performance of the Endoscopic Cap Electrode (ECE50)
Acronym: ECE50
Status: Active, not recruiting | Type: Observational
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021REG002
Record Dates: First submitted 2021-12-22; First posted 2022-02-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Vocal Fold Paresis; Laryngeal Dystonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this registry is to confirm the safety and the performance of the ECE50 in medical routine by collecting data.

DETAILED DESCRIPTION:
The Endoscopic Cap Electrode (ECE50) has been designed for the delivery of electrostimulation to selected laryngeal muscles. The primary objective of this registry is to retrieve real-life data on the safety and performance of the Endoscopic Cap in medical routine. Subject's participation will last a maximum of 2 hours. Upon successful conclusion of the screening session starts the testing session of the ECE50. The ECE50 has been designed to be placed on the top of a videoendoscope for the delivery of electrostimulation to the laryngeal region. The stimulation and reaction of the muscles can provide information about the presence and type of dysfunctions and thus influence the treatment procedure. Being a registry a collection of records generated within routine medical procedures with a medical device approved for the EU market, it does not pose additional risks for the patients participating in it.

ELIGIBILITY:
Inclusion Criteria:

* Legal adults (i.e., as a general rule patients ≥ 18 years old)
* Legal adults requiring a diagnosis for a disorder that could be traced back to uni- or bilateral dysfunction of one or more laryngeal muscle(s) of the posterior cricoid region
* Signed and dated informed consent before the start of any registry-specific procedure for all the recruited subjects

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* Use of an active medical implant
* Known allergies or intolerance to the material used for this registry
* Parallel participation in a device/drug registry in the period of data collection, which could confound the results of the registry
* Anything that, in the opinion of the Registry Responsible, would place the subject at increased risk or preclude the subject's full compliance with the general requirements of this registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Target population: adults of both sexes who, in the expert opinion of the registry responsible is in need of an ECE50 examination
  * Accessible population: target population matching the selection criteria
  * Intended population: accessible population that can be recruited by the registry sites
  * Actual population: intended population who signed the ICF
  * Analytic population: actual population compatible with PP analysis
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2021-12-16 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2031-12-16 (Estimated)

PRIMARY OUTCOMES:
Confirm the safety | Immediately after the intervention
  Adverse event report analysis
Assess the performance of the ECE50 | During the intervention
  Comparison between the result of the ECE50 stimulation, Laryngeal Electromyography (LEMG), videolaryngoscopy

SECONDARY OUTCOMES:
Standardize the medical procedure for the ECE50 | Immediately after the intervention
  Descriptive evaluation of the ECE50 stimulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Berit Schneider-Stickler, Prof.Dr.med., Principal Investigator — Univ. Klinik für Hals-, Nasen- und Ohrenkrankheiten, Vienna
Locations (1):
- Univ. Klinik für Hals-, Nasen- und Ohrenkrankheiten, Vienna, Austria